CLINICAL TRIAL: NCT06255912
Title: A Phase II Clinical Trial Assessing the Safety, Tolerability, and Pharmacokinetics of LTC004 in Combination With MIL-97 ± Chemotherapy in Patients With Advanced or Metastatic Pancreatic Cancer
Brief Title: Clinical Trial for Advanced or Metastatic Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, NING LI, professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LTC004-201
Record Dates: First submitted 2023-12-26; First posted 2024-02-13 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTC004 + MIL-97 (Experimental)
  Interventions: Drug: LTC004 + MIL-97
- LTC004 + MIL-97+ chemotherapy (Experimental)
  Interventions: Drug: LTC004 + MIL-97+chemotherapy

INTERVENTIONS:
Drug: LTC004 + MIL-97 — Dose group 1：MIL97:0.2mg/kg,Day1,Q3W,LTC004:90ug/kg,Day3,Q3W Dose group 2:MIL97:0.2mg/kg,Day1,Q3W,LTC004:180ug/kg,Day3,Q3W Dose group -1:MIL97:0.2mg/kg,Day1,Q3W,LTC004:45ug/kg,Day3,Q3W
  Arms: LTC004 + MIL-97
Drug: LTC004 + MIL-97+chemotherapy — LTC004 + MIL-97+chemotherapy
  Arms: LTC004 + MIL-97+ chemotherapy

SUMMARY:
This is a Phase II clinical trial assessing the safety, tolerability, and pharmacokinetics of LTC004 in combination with MIL-97 ± chemotherapy in patients with advanced or metastatic pancreatic cancer.

This experiment is divided into two parts: the dose increasing stage (stage 1) and the dose expanding stage (stage 2). For those enrolled in the planned expansion phase, the dose should have passed the safety assessment during the dose escalation phase.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign the informed consent form
2. Patients with inoperable advanced pancreatic cancer who have experienced progression during or after receiving at least one systemic treatment line, including the modified FOLFIRINOX regimen, capecitabine and/or gemcitabine, erlotinib, with or without platinum agents (oxaliplatin, cisplatin, or carboplatin), or taxane agents (paclitaxel, nab-paclitaxel, or docetaxel), etc.; patients with documented first recurrence after adjuvant therapy can also be included in this study.
3. Diagnosed histologically or cytologically as pancreatic ductal adenocarcinoma
4. During screening, at least one measurable tumor lesion must be present (according to RECIST v1.1 criteria).
5. During screening, the Eastern Cooperative Oncology Group (ECOG) performance status should be ≤1.
6. During screening, an expected survival of ≥12 weeks is required, along with good organ function
7. Before the initial administration of the investigational drug, systemic chemotherapy should have been completed for at least 4 weeks, monoclonal antibody therapy for at least 4 weeks, small molecule targeted therapy for at least 2 weeks, or for at least 5 half-lives of the drug (whichever is longer). Additionally, treatment with domestically approved anti-tumor Chinese herbal medicine or traditional Chinese medicine with anti-tumor effects should have been completed for at least 2 weeks according to the National Medical Products Administration (NMPA).
8. Non-fertile female patients, or fertile female patients with a negative pregnancy test result, who commit to using effective contraception or practicing abstinence from the screening period until 6 months after the last dose of the investigational drug (see Appendix V). Similarly, male patients commit to using effective contraception or practicing abstinence from the screening period until 6 months after the last dose of the investigational drug.
9. Understand and voluntarily sign the written Informed Consent Form (ICF), willing and able to complete regular visits, follow the treatment plan, undergo laboratory tests, and participate in other trial procedures.

Exclusion Criteria:

1. Severe history of allergic reactions to other monoclonal antibodies or fusion protein medications.
2. Previous treatments including any immunotherapies such as immune checkpoint inhibitors, CD40, etc.
3. Untreated, unstable, or uncontrolled central nervous system (CNS) metastases, except for cases where: within at least 4 weeks before initial dosing, clinical MRI scans demonstrate disease stability (at least 2 consecutive scans within 6 months before enrollment, including one scan within 28 days before screening) and no progression or uncontrolled neurological symptoms or signs (such as seizures, headaches, central nausea, vomiting, progressive neurological deficits, papilledema).
4. Uncontrolled pleural effusion, pericardial effusion, or ascites as determined by the investigator (requiring repeated drainage, multiple times per month, or more frequently).
5. Patients with untreated or clinically symptomatic spinal cord compression that has not been controlled (except for cases where patients have been treated and symptoms have stabilized, imaging shows stability for at least 4 weeks before initial dosing, without evidence of brain edema, and no need for corticosteroid treatment).
6. Having had ≥2 malignancies within 5 years before the initial dosing. Exceptions include cured early-stage malignancies (carcinoma in situ or stage I tumors), such as adequately treated cervical carcinoma in situ, thyroid cancer, basal cell or squamous cell skin carcinoma.
7. Resting moderate to severe dyspnea due to advanced cancer or its complications, severe primary lung diseases, current requirement for continuous oxygen therapy, or clinically active interstitial lung disease (ILD) or pneumonia.
8. Having experienced grade ≥3 interstitial pneumonia during previous anticancer treatment.
9. Individuals with active pulmonary tuberculosis infection within the year prior to enrollment as identified by medical history or screening examinations, or those with a history of active pulmonary tuberculosis infection more than one year ago but have not received proper treatment
10. Severe infections within the first four weeks before the initial medication, including but not limited to septicemia requiring hospitalization, severe pneumonia, etc.; Active infections of CTCAE ≥2 grade requiring systemic antibiotic treatment within two weeks before the initial medication
11. A history of severe cardiovascular diseases, including but not limited to severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, second or third-degree atrioventricular block, etc.; Occurrence of acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or above cardiovascular events within six months before the initial medication; New York Heart Association (NYHA) functional class II or left ventricular ejection fraction (LVEF) < or clinically uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg)
12. During screening, patients with active hepatitis B (Hepatitis B virus titers > lower limit of detection) or hepatitis C. Patients positive for Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) can participate in this study if the Hepatitis B virus (HBV) deoxyribonucleic acid (DNA) test is below the upper limit of normal detection at the respective research center. Patients positive for Hepatitis C virus (HCV) antibodies can participate in this study if the HCV ribonucleic acid (RNA) test is below the upper limit of normal detection at the respective research center
13. Patients who test positive for syphilis during screening; Patients with active or previously experienced and potentially relapsing autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis), except for clinically stable patients with autoimmune thyroid disease; Those with immunodeficiency diseases or a history thereof, including positive serum testing for human immunodeficiency virus (HIV); Individuals who have experienced significant clinically relevant bleeding symptoms within 3 months before the first administration.
14. Patients who received systemic immunosuppressive therapy within 2 weeks before the first dose (including but not limited to glucocorticoids, cyclophosphamide, azathioprine, methotrexate, or thalidomide);
15. Those who have used immune modulators within 2 weeks before the first dose (or 5 half-lives of the drug, whichever is longer), including but not limited to thymopentin, IL-2, IL-15, interferons, etc.;
16. Patients who underwent curative radiotherapy within 4 weeks before the first dose, and those who received palliative radiation within 14 days before the first dose;
17. Patients with tumors invading vital surrounding organs (such as the aorta and trachea), or with a risk of esophageal or tracheal fistula, or esophageal pleural fistula; 18. Individuals with a history of gastrointestinal perforation or fistula within 6 months before the first dose;

19.Patients who received other investigational drugs or treatments not yet approved within 4 weeks before the first dose.

20.Subjects who have received live attenuated vaccines or live vaccines within 4 weeks before the first dose, or are expected to receive live attenuated vaccines or live vaccines during the study period; 21.Individuals who underwent major surgery within 4 weeks before the first dose (excluding diagnostic procedures), are expected to undergo major surgery during the study period (excluding diagnostic procedures), or have had diagnostic or minimally invasive surgery within 7 days before the first dose (excluding puncture biopsies); 22. Patients whose adverse reactions from previous anticancer therapy have not recovered to Grade 1 according to CTCAE 5.0 (except for Grade 2 alopecia and Grade 2 neuropathy caused by chemotherapy, Grade 2 hypothyroidism induced by anticancer therapy, and Grade 2 reduction in hemoglobin); 23.Individuals who have previously undergone allogeneic hematopoietic stem cell transplantation or solid organ transplantation; 24.Pregnant or lactating women; 25.Subjects judged by the investigator to have a history of other serious systemic diseases or any other reasons (such as mental illness, alcoholism, substance abuse, or drug abuse) that may affect trial compliance and make them unsuitable for participation in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | within 3 weeks
  safety
Maximum tolerated dose Tolerated Dose Dose | during treatment（through study completion, an average of 1 year）
  Maximum tolerated dose
Treatment Emergent Adverse Events | during treatment（through study completion, an average of 1 year）
  safety

SECONDARY OUTCOMES:
overall response rate | At the end of every 2 cycles(each cycle is 21 days）
  efficacy